CLINICAL TRIAL: NCT02380664
Title: Swimming Training Repercussion on Metabolic and Structural Bone Development; Benefits of the Incorporation of Whole Body Vibration or Plyometric Training. The RENACIMIENTO Project
Brief Title: Swimming Training Repercussion on Metabolic and Structural Bone Development; Benefits of the Incorporation of Whole Body Vibration or Plyometric Training: The RENACIMIENTO Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, German Vicente-Rodríguez, Lecturer, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEP2011-29093
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Body Composition
Keywords: swimmers; adolescent swimmers; whole-body vibration; bone and bones; body composition

ARMS (4):
- Swimmers (No Intervention): Swimmers that continue their normal swimming activity
- WBV swimmers (Experimental): Swimmers that perform a whole-body vibration training
  Interventions: Device: Whole-body vibration (Powerplate®)
- Plyometric swimmers (Experimental): Swimmers that perform a plyometric training
  Interventions: Behavioral: Jumping intervention
- Sedentary controls (No Intervention): Controls that do not perform swimming or other physical activities

INTERVENTIONS:
Device: Whole-body vibration (Powerplate®) — Swimmers will perform a 15 minute whole-body vibration training 3 times per week. This intervention will be performed with a Powerplate®. The vibration protocol will be progressive starting with 30 Hz and an amplitude op 4 mm reaching at the end of the protocol 38 Hz and 4 mm amplitude.
  Arms: WBV swimmers
Behavioral: Jumping intervention — Swimmers will perform a jumping intervention, 15 minutes 3 times per week. Jumps will include drop jumps, one leg jumps, squat jumps and countermovement jumps.
  Arms: Plyometric swimmers

SUMMARY:
Swimming training is associated with decreased bone mass and lower bone mass acquisition during growth periods, mainly when compared to other weight-bearing sports. Little information is available in adolescents pointing in the same direction but still controversial.

On the other hand, bone strength do not only depends on bone mass but on bone structure and microarchitecture. The cross sectional area, cortex thickness or trabecular density are important aspects of bone health. There are few studies on the effect of swimming on bone architecture of adolescents. This information is relevant for present and future health of adolescents practicing swimming and for all the organizations promoting this sport. Jumping and whole body vibration training programs seem to elicit important osteogenic effects; however, there is little information on this regard in adolescent population, even less in these adolescents with potentially decreased bone acquisition such as swimmers.

The main aims of this research project are therefore, to analyze the effect of swimming training on bone mass, metabolism, structure and architecture in adolescents analyzing possible relationships among them. Secondly, to test whether including short boots of jumping or whole body vibration may be able to palliate the possible deleterious effects of swimming and facilitate a normal or even healthier bone development. And finally to study the durability of training-related bone gains over time.

ELIGIBILITY:
Inclusion Criteria:

* Specific for the swimmers: With a history of training at least 3 years for more than 6 hours per week and currently still training
* Specific for the control group: Subjects that do not perform more than 3 hours of physical activity per week

Exclusion Criteria:

* Non-caucasian
* Smoking
* Taking medication affecting bone

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in body composition during 3 years evaluated by dual energy X-ray | Change from baseline in body composition at 3 years

SECONDARY OUTCOMES:
Change in bone strength and structure evaluated by peripheral quantitative computed tomography | Change from baseline in bone strength and structure at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: German Vicente-Rodríguez, PhD, Principal Investigator — GENUD Research Group, Universidad de Zaragoza, Spain